CLINICAL TRIAL: NCT07134816
Title: Cost-utility Study of Cognitive-behavioral Management of Auditory Hallucinations in Schizophrenic Disorder
Acronym: VOICES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other); Centre Hospitalier Universitaire de Nîmes (Unknown); Centre Hospitalier de Béziers (Unknown); University Hospital, Clermont-Ferrand (Other); Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL22_0337
Record Dates: First submitted 2025-02-04; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Auditory Hallucinations; Schizophrenia Spectrum
Keywords: Cognitive Behavioral Therapy; Non Pharmacological Intervention (NPI); cost utility study
MeSH Terms: conditions — Hallucinations | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To limit classification bias, hetero-questionnaires and collection of clinical endpoints will be collected by an assessor blinded to the study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive and behavioral therapy for auditory hallucinations (Experimental)
  Interventions: Other: Cognitive and behavioral therapy for auditory hallucinations
- Usual treatment (Active Comparator)
  Interventions: Other: Usual treatment

INTERVENTIONS:
Other: Cognitive and behavioral therapy for auditory hallucinations — Consists of 16 one-hour individual sessions (one session per week over a 16-week period) of cognitive behavioral therapy, divided into three types of interventions (modules) that have been independently proven to be effective in the management of auditory hallucinations.
  Arms: Cognitive and behavioral therapy for auditory hallucinations
Other: Usual treatment — Consists of an antipsychotic medication treatment (including dosage changes and molecule changes.), regular consultation with a psychiatrist (once a month on average), and if necessary, one-off psychological support or family interventions not including specific CBT for positive symptoms
  Arms: Usual treatment

SUMMARY:
The aim of the study is to assess the effectiveness and costs of a cognitive-behavioral treatment (CBT) for auditory hallucinations (psychotherapy) as an adjunct to usual care, comparing it to the effectiveness and costs of usual care alone. Usual care is defined as the use of medication, regular consultations with your psychiatrist, and, if necessary, day hospital care.

The study plans to include 240 participants across several hospitals in France (multicenter study). Each participant will be randomly assigned to either the intervention group (cognitive-behavioral therapy) or the control group (usual treatment). Participants assigned to the control group will have the opportunity to receive therapy for auditory verbal hallucinations (AVHs) after the study.

After an initial inclusion assessment (V0), the participant will be randomly assigned to one of the two groups after the V1 assessment. Additional evaluations will be conducted after inclusion at 4 months, 8 months, and 12 months.The evaluations consist of questionnaires to assess intensity and severity of AVHs / beliefs related to AVHs, clinical status, well-being, depression, suicidal thoughts, quality of life, functioning (mobility/autonomy/pain, etc.), sleep and costs related to care.

At Visit 1, after obtaining consent for participation in the study on behalf of your ward, the investigator will also collect their social security number, full date of birth, and gender, which will allow us to gather information on actual healthcare consumption from the healthcare system.

The VOICES intervention will consist of 16 one-hour individual sessions (one session per week over a 16-week period), divided into several types of intervention (modules) that have been independently proven to treat AVHs. The VOICES intervention is modular, personalized, and incorporates patient preference. Following an initial clinical assessment, patients will be offered first the GIVE intervention (8 sessions) and subsequently a choice of treatment modules, delivered by a clinical psychologist.

After this first module (GiVE Intervention), three other intervention modules will be proposed. These three additional modules comprise seven sessions each. One additional relapse prevention sessions will be scheduled at the end of these modules.

- The GiVE intervention is divided into five modules: (1) Coping - exploring ways to manage voices; (2) Me - targeting negative beliefs about the self; (3) My Voices - targeting unhelpful beliefs about voices; (4) My Relationships - improving assertiveness in difficult relationships; and (5) Looking to the Future - making plans to continue the use of new skills. Modules 2, 3 and 4 were each offered over two sessions (six sessions in total), and modules 1 and 5 were each one session long.

After the GivE intervention three modules will be offered will be :

* "Relating CBT" is based on a large body of research which has shown that voice hearers personify their voices and establish relationships with them, which largely correspond to the relationships they generally establish with the people around them. The aim of relational therapy will be to modify this relationship and enable the voice hearer to develop assertive and balanced behaviours towards them.
* The individual "Mindfulness Program for Voices" will be delivered individually and will include guided mindfulness exercises, complemented by discussions aimed at cultivating mindful responses as alternatives to automatic or habitual reactions.

  * Imagery rescripting for distressing voices will consist of a series of targeted imagery-based interventions guided by a micro-formulation approach. This method will focus on the identification and transformation of discrete, emotionally salient mental images linked to specif distressing experiences

All participants will receive medical monitoring, and the treatment will be the same in both groups. No treatment will be prohibited if deemed necessary for your health. At any time, participants have the right to withdraw their consent and stop participating in the research, without any change to their care, as long as the patient's condition does not require otherwise.

The expected benefits for participants are a significant improvement in the symptoms as well as psychosocial functioning, leading to greater autonomy in daily life and an improved quality of life. In the control group, the follow-up will likely be more attentive than usual, with regular evaluations. In any case, there is no loss of opportunity for the participant regardless of the group assignment. Additionally, random assignment to the control group allows participants to benefit from AVH therapy after the study.

When the research is completed, participants will be informed of the overall results by the investigator as soon as they are available, if wished.

Participation in this research will not incur any additional costs compared to the usual follow-up for this condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenic disorder according to DSM 5 as assessed by the investigating psychiatrist during the screening medical examination
* Age between 15 and 45 years inclusive
* Patients hearing AVHs for at least 3 months
* Patient with a score of at least 2 on the distress intensity item of the hallucinations subscale of the Psychotic Symptom Rating Scale (PSYRATS-AH).

Exclusion Criteria :

* Patients hospitalized full-time for acute decompensation of their schizophrenic disorder
* Patients with a history of severe head trauma and/or neurological pathology with cognitive impact
* Patients with a characterized depressive state (Calgary scale score>9)
* Patients unable to understand, speak and read French
* Patients with moderate to severe intellectual disability (pre-morbid IQ estimated by fNART<70)
* Hallucinations of organic or toxic origin
* Suicidal ideation type 4 or 5
* Pregnant and breastfeeding women
* Main diagnosis of substance abuse or dependence, having received full CBT care (minimum 16 hours) for psychotic symptoms in the past year
* Participation in another interventional study in which the patient benefits from psychological intervention
* Patient unable to give written informed consent, for minors, absence of signatures of the legal representative(s), for adults patients benefiting from guardianship, absence of written consent from the guardian, for patients under curatorship, failure to inform the curator, for patients in psychiatric care at the request of a third party, absence of consent from the trusted person
* Not able to carry out all visits and follow the study procedures
* Not affiliated or beneficiary of a social security scheme

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incremental cost-utility ratio | Baseline, 4 months, 8 months, 12 months
  Incremental cost-utility ratio (ICUR) at 12 months, of the management of auditory hallucinations by CBT compared to usual treatment. The preferred outcome criterion is the QALY (Quality Adjusted Life Years) unit of measurement of the duration of life weighted by the quality of life related to health (HAS 2020), calculated from the utilities derived from the EuroQuality of life 5 dimensions questionnaire (EQ5D-5L).

SECONDARY OUTCOMES:
Distress associated with AVHs and frequency | Baseline, for intervention group 6 weeks to 11 weeks, 4 months, 8 months, 12 months
  Using the Psychotic Symptom Rating Scales - Auditory Hallucinations (PSYRATS-AH; Haddock et al., 1999; Favrod et al., 2012 for French validation), a hetero-questionnaire consisting of 11 items designed to measure the severity of various dimensions of the auditory hallucination experience. The items are grouped into four factors: distress (negative content, distress, and control), frequency (frequency, duration, and disruption), attribution (location and origin of the auditory hallucinations), and intensity of sound. Each item is rated on a scale from 0 ("not at all") to 4 ("always"). The total score ranges from 0 to 44.
Beliefs about voices | Baseline, months 4, 8 and 12
  Using The Beliefs About Voices Questionnaire (BAVQ-R, Chadwick and al, 2000) a self-report questionnaire that assesses beliefs, emotional, and behavioral consequences related to auditory hallucinations (AHs). It initially contains 35 items, each rated from 0 ("strongly disagree") to 3 ("strongly agree"), and is divided into 5 subscales: Power, Malevolence, Benevolence, Resistance, and Engagement. We will consider the total score for the four subscales: Power, Malevolence, Resistance, and Engagement (total score ranging from 0 to 12).
Maastricht Semi-structured Interview | Baseline only for The Maastricht interview
  The Maastricht Semi-structured Interview, developed by Romme and Escher (2000), is a precursor to the early work on the experience of AVHs in the Netherlands. It allows for the assessment of this phenomenological experience through a variety of individual variables such as intensity, volume, and number of AVHs, while also addressing the individual's environmental spheres and potential journey through different psychiatric care services.
Auditory Hallucination Rating Scale | Baseline, months 4, 8 and 12
  Auditory Hallucination Rating Scale (AHRS), French validation by Dondé et al., 2020. This scale includes 7 questions regarding the frequency, intensity, or intentional valence of AVHs.
Hallucination Relationship Scale | Baseline, months 4, 8 and 12
  Hallucination Relationship Scale (Approve Questionnaire, Hayward et al., 2020). This scale consists of 30 items measuring both assertiveness in relation to AVHs and assertiveness in everyday life in human relationships.
Assessment of psychotic symptomatology | Baseline, 4, 8, 12 months
  For the psychotic symptoms, the "Positive And Negative Syndrome Scale" (PANSS): The PANSS is a 30-item hetero-assessment scale, rated from 1 to 7, which measures the symptomatology specific to psychotic disorders, particularly schizophrenic disorders. It calculates scores for 3 syndromic dimensions: positive (7 items), negative (7 items), and general psychopathology (16 items), from both a categorical and dimensional perspective.
Psychiatric comorbidities | Baseline
  For the comorbidities,the "Mini International Neuropsychiatric Interview" (M.I.N.I) is a structured diagnostic interview, with a short duration (approximately 20 minutes) exploring in a standardized way, the main psychiatric disorders according to the DSM IV. The M.I.N.I version 5.0 is divided into identified modules, each corresponding to a diagnostic category. We will use modules A, D, E, F, G, H, I, M, N, O.
Depression assessment | Baseline, 4 months, 8 months, 12 months
  Calgary Depression Scale for Schizophrenia (CDSS, Addington & Addington, 1990). This scale is designed to assess depression in individuals with schizophrenia. The questionnaire consists of 9 items (depressed mood, despair, self-deprecation, reference ideas with a theme of guilt, pathological guilt, morning depression, early awakening, suicidal thoughts, and observed depression) covering the past two weeks. Each item is rated on a 4-point Likert scale ranging from: "Absent" (0) to "Severe" (3). The total score is obtained by adding the items and provides a score out of 27.
Suicidal risk | Baseline, 4, 8 and 12 months
  Columbia Suicide Severity Rating Scale (C-SSRS, Posner et al., 2011). The C-SSRS measures four dimensions. The first is the severity of suicidal ideation, which is assessed on a 5-point ordinal scale. The second is the subscale of intensity of suicidal thoughts, which includes 5 items, each rated on a 5-point ordinal scale: frequency, duration, controllability, deterrents, and reason for ideation. The third is the behavioral subscale, assessed on a nominal scale, which includes actual, aborted, and interrupted attempts, preparatory behavior, and non-suicidal self-injury. The fourth is the lethality subscale, which evaluates actual attempts; actual lethality is rated on a 6-point ordinal scale. Suicidal risk is ultimately determined by the clinician's judgment when administering the scale.
Psychological well-being | Baseline, 4, 8 and 12 months
  PERMA Psychological Well-Being Scale (Seligman, 2011). This scale consists of 10 items encompassing four factors: positive emotion, relationships, having a sense of purpose in life, and personal accomplishment. Each question is rated on an 11-point Likert scale, ranging from "0 = never" to "10 = always," "0 = not at all" to "10 = completely," or "0 = very poor" to "10 = excellent," depending on the content of the question.
EQ-5D-5L (EuroQol) | Baseline, 4 months, 8 months, 12 months
  The EQ-5D-5L (EuroQol) is a multi-attribute health status classification system consisting of 5 attributes: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D-5L will be used to measure the effectiveness of the innovation in terms of QALYs (Quality-Adjusted Life Years), which is an which is an indicator where health states are weighted by quality of life.
The Global Assessment of Functioning | Baseline, 4 months, 8 months, 12 months
  The Global Assessment of Functioning (GAF) is a numerical scale (ranging from 0 to 100) used in psychiatry to assess an individual's psychological, social, and occupational functioning.
Functional Remission of General Schizophrenia | Baseline, 4 months, 8 months, 12 months
  The Functional Remission of General Schizophrenia (FROGS) scale will be used to assess patients' functioning (Llorca et al., 2009).
Estimation of premorbid IQ | Baseline, months 4, 8 and 12
  Premorbid IQ by the fNART (French version of the National Adult Reading Test, Mackinnon & Mulligan (2005)). The ƒNART is based on the ability to pronounce 40 words with irregular spelling. It offers clinicians and researchers an easy method of estimating premorbid intelligence using a robust test in the face of cognitive decline.
Sleep assessment | Months 8 and 12
  Using the Insomnia Severity Index (ISI), developed to assess the severity of insomnia complaints and their daytime repercussions on daily activities. The first item evaluates the intensity of insomnia complaints such as difficulty falling asleep, maintaining sleep, and early awakening, each separately. One item assesses the overall satisfaction of the subject with their sleep, and another item evaluates concerns about insomnia. Finally, two items assess the impact on daily activities. Each item is rated by the patient on a scale from 0 to 4. The total score is obtained by adding the scores for each item. The total score ranges from 0 to 28.
Medication Adherence Rating Scale | Baseline, 4, 8 and 12 months
  The "Medication Adherence Rating Scale" (MARS) will assess adherence to medication treatment. This is a self-administered questionnaire of 10 items, yes/no answer

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, Montpellier, Occitanie, France

IPD SHARING:
Plan to Share IPD: Undecided